CLINICAL TRIAL: NCT03952026
Title: Impact of Associated Abdominal Injuries on Clinical and Operative Outcome in Pelvic Fractures - a Multicenter Study From the German Pelvic Registry
Brief Title: Impact of Associated Abdominal Injuries on Clinical and Operative Outcome in Pelvic Injuries
Status: Completed | Type: Observational
Sponsor: BG Trauma Center Tuebingen (Other)
Responsible Party: Principal Investigator, Markus Küper, Principal Investigator, BG Trauma Center Tuebingen
Other Study IDs: 001
Record Dates: First submitted 2019-05-11; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Pelvic Ring Fracture; Acetabular Fracture; Abdominal Trauma; Polytrauma
Keywords: Pelvic trauma; Pelvic ring fracture; Acetabular Fracture; Abdominal Trauma; Polytrauma; Reduction quality
MeSH Terms: conditions — Abdominal Injuries; Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- isolated pelvic fracture: Patients with an isolated pelvic fracture
  Interventions: Procedure: osteosynthesis of the pelvis
- combined abodominal/pelvic injury: Patients with a combined injury of a pelvic fracture and an abdominal injury.
  Interventions: Procedure: osteosynthesis of the pelvis

INTERVENTIONS:
Procedure: osteosynthesis of the pelvis — Osteosynthetic Fixation of the pelvic fracture

SUMMARY:
Pelvic fractures are severe injuries which require advanced orthopedic surgical skills to treat. On the other hand, abdominal injuries are severe injuries, which might require quick general surgical treatment. The combination of both injuries is a challenge for orthopedic surgeons, as the abdominal injury might lead to a delayed surgical treatment of the pelvic fracture. Whether an associated abdominal injury influences the quality of care of pelvic fractures, is aim of this registry study.

DETAILED DESCRIPTION:
The German Pelvic Registry of the German Trauma Society is a multicenter prospective registry which collects data of patients with pelvic injuries since 2003. Beside demographic data (including concomitant injuries) allowing for epidemiological evaluations of the development of surgical care in these patients, namely the operative care is focus of this registry. Beside the chosen procedure or surgical approach, this includes both intraoperative data like time until operation, duration of the procedure or intraoperative blood loss and reduction parameters (pre- and postoperative fracture steps). The clinical course is recorded also including overall morbidity, overall mortality and osteosynthesis-related complications.

The influence of a concomitant abdominal trauma on the quality of care regarding operative parameters like reduction quality or the clinical course in pelvic injuries has not been investigated yet.

The investigators therefore retrospectively analyze the prospective consecutive data of patients from the multicenter German Pelvic Registry of the German Trauma Society in the years 2003 - 2017. Demographic, clinical and operative parameter were recorded and compared in two groups (isolated pelvic fracture vs. combined abdominal/pelvic trauma).

ELIGIBILITY:
Inclusion Criteria:

* Pelvic fracture

Exclusion Criteria:

* no agreement to participate in the registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a pelvic fracture Group 1: isolated pelvic fracture Group 2: combined abdominal/pelvic injury
Sampling Method: Non-Probability Sample
Enrollment: 16359 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
"Matta" Grading | through study completion, at least 1 year after inclusion
  Quality of the reduction of the pelvic fracture measured in mm residual step at the fracture's site. A residual step of 0-2mm is graded as an "anatomical reduction" (=Matta 1), a residual step of 2-3mm is graded as an "Imperfect reduction" (=Matta 2) and a residual step >3mm is graded as a "poor reduction" (=Matta 3).
Overall morbidity | through study completion, at least 1 year after inclusion
  Rate of overall complications

SECONDARY OUTCOMES:
osteosynthesis-associated complications | through study completion, at least 1 year after inclusion
  Rate of osteosynthesis-associated complications
length of hospital stay | through study completion, at least 1 year after inclusion
  Duration of the inpatient Treatment, measured in days.
Time until definitive pelvic surgery | through study completion, at least 1 year after inclusion
  The time until the definitive surgical procedure for the pelvic fracture, measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Markus A Küper, MD, Principal Investigator — BG Trauma Center Tübingen
Locations (1):
- BG Trauma Center, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Kuper MA, Bachmann R, Wenig GF, Ziegler P, Trulson A, Trulson IM, Minarski C, Ladurner R, Stockle U, Hoch A, Herath SC, Stuby FM; Working Group on Pelvic Fractures of the German Trauma Society. Associated abdominal injuries do not influence quality of care in pelvic fractures-a multicenter cohort study from the German Pelvic Registry. World J Emerg Surg. 2020 Jan 17;15:8. doi: 10.1186/s13017-020-0290-x. eCollection 2020. PMID 31988652